CLINICAL TRIAL: NCT01872260
Title: A Phase Ib/II, Multicenter Study of the Combination of LEE011 and BYL719 With Letrozole in Adult Patients With Advanced ER+ Breast Cancer
Brief Title: Study of LEE011, BYL719 and Letrozole in Advanced ER+ Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2107; 2023-509511-84-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT05038631 (Available)
Record Dates: First submitted 2013-05-30; First posted 2013-06-07 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Hormone-receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LEE011 + letrozole Arm 1 (Experimental): LEE011 - 28 day cycles (21 days followed by a 7 day break - dose escalating), letrozole - 2.5 mg/day
  Interventions: Drug: LEE011; Drug: Letrozole
- BYL719 + letrozole Arm 2 (Experimental): BYL719 - daily (dose escalating) letrozole - 2.5 mg/day
  Interventions: Drug: Letrozole; Drug: BYL719
- LEE011 + BYL719 + letrozole Arm 3 (Experimental): LEE011 - 28 day cycles (21 days followed by a 7 day break -dose escalating), BYL719 - daily (dose escalating), letrozole 2.5 mg/day
  Interventions: Drug: LEE011; Drug: Letrozole; Drug: BYL719
- LEE011+ BYL719+letrozole Arm 4 (Experimental): LEE011-daily (dose escalating), BYL719 -daily (dose escalating), letrozole 2.5 mg/day
  Interventions: Drug: LEE011; Drug: Letrozole; Drug: BYL719

INTERVENTIONS:
Drug: LEE011 — LEE011 - 28 day cycles (21 days followed by a 7 day break) for Arms 1, 3. LEE011 28 days cycles (continuous) Arm 4.
  Arms: LEE011 + BYL719 + letrozole Arm 3; LEE011 + letrozole Arm 1; LEE011+ BYL719+letrozole Arm 4
Drug: Letrozole — Letrozole 2.5 mg/day
Drug: BYL719 — BYL719 - 28 days cycle (continuous) for Arm 2; 3 and 4
  Arms: BYL719 + letrozole Arm 2; LEE011 + BYL719 + letrozole Arm 3; LEE011+ BYL719+letrozole Arm 4

SUMMARY:
The purpose of this trial is to inform the future clinical development of the two investigational agents in ER+ breast cancer, LEE011 (CDK4/6 inhibitor) and BYL719 (PI3K-alpha inhibitor).

This is a multi-center, open-label Phase Ib study. The Phase Ib dose escalation will estimate the MTD and/or RP2D for three regimens: two double combinations, LEE011 with letrozole and BYL719 with letrozole, followed by triple combinations of LEE011 + BYL719 with letrozole (Arms 3 and 4).

The Phase Ib dose escalation part will be followed by Phase Ib dose expansions to further characterize the safety, tolerability, PK and preliminary clinical anti-tumor activity of the combinations. Optional crossover for patients who have progressed while on dose escalation or dose expansion with doublet treatment on Arms 1 or 2 to be treated with the triplet combination (Arm 3) after the determination of the RP2D for Arm 3; is no longer permitted after protocol amendment 6.

Approximately 270 adult women with ER+/HER2- locally advanced or metastatic breast cancer will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, Estrogen-receptor positive and/or Progesterone-receptor positive breast cancer
* Phase Ib dose escalation only: Any number of prior lines of endocrine therapy is allowed with the exception of cytotoxic therapy which is limited to one prior line administered in the advanced (metastatic or locally advanced) setting.
* Phase Ib dose expansions Arms 1, 2 and 3
* No prior systemic treatment in the advanced (metastatic or locally advanced) setting with the exception of treatment with letrozole for a maximum of one month prior to starting study treatment.
* Patients who received (neo)adjuvant therapy for breast cancer are eligible. Prior therapy with letrozole or anastrozole in the (neo)adjuvant setting is permitted if the disease-free interval is greater than 12 months from the completion of treatment.

Exclusion Criteria:

* HER2-overexpression in the patient's tumor tissue
* Patients with active CNS or other brain metastases
* Major surgery within 2 weeks
* Acute or chronic pancreatitis
* Bilateral diffuse lymphangitic carcinomatosis
* Another malignancy within 3 years
* Receiving hormone replacement therapy that cannot be discontinued
* Impaired cardiac function
* Patients with clinically manifest diabetes mellitus (treated and/or clinical signs or with fasting glucose ≥ 126 mg/dL / 7.0 mmol/L or hemoglobin A1c >6.5%), history of gestational diabetes mellitus or documented steroid-induced diabetes mellitus.
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities (DLTs) - Phase lb only | 28 days
Safety and tolerability | Average 18 months
  Adverse Events (AEs), serious AEs (SAEs), changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs), dose interruptions, reductions and dose intensity.
PK profiles of LEE011 and letrozole | 18 months
  To characterize PK profiles of LEE011 and Letrozole.

SECONDARY OUTCOMES:
Safety and tolerability of LEE011 in combination with letrozole, BYL719 in combination with letrozole, and the triple combination of LEE011 +BYL719 with letrozole | Average 24 months
  Safety and tolerability will be determined by type, frequency and severity of adverse events and laboratory abnormalities per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Plasma concentration-time profiles of LEE011, BYL719 and letrozole | Average 24 months
  To characterize the PK profiles of LEE011, BYL719, and letrozole when used in combination as well as to evaluate any other clinically significant metabolites that may be identified.
Overall Response Rate (ORR) | Average 24 months
  ORR is defined as the proportion of patients with a best overall response of complete response or partial response.
Duration of Response (DOR) | Average 24 months
  DOR is calculated as the time from the date of first documented response (complete response (CR) or partial response (PR)) to the first documented date of progression or death due to underlying cancer.
Progression Free Survival (PFS) | Average 24 months
  PFS is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause.
Pharmacokinetics (PK) parameters, including but not limited to AUCtau, Cmin, Cmax, Tmax, accumulation ratio (Racc) | Average 24 months
  To characterize the PK profiles of LEE011, BYL719, and letrozole when used in combination as well as to evaluate any other clinically significant metabolites that may be identified.
Safety and tolerability of the triple combination of LEE011 +BYL719 with letrozole in patients previously treated with either doublet | Average 24 months
  Safety and tolerability will be determined by type, frequency and severity of adverse events and laboratory abnormalities per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (10):
  - Univ of California at San Diego Moores Cancer Ctr, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Massachusetts General Hospital SC-5, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Ctr, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Mays Cancer Ctr Uthsa Mdacc, San Antonio, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (3):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain
- Novartis Investigative Site, Pisa, PI, Italy
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (3):
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Bellinzona, Switzerland
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ji Y, Yartsev V, Quinlan M, Serra P, Wang Y, Chakraborty A, Miller M. Justifying Ribociclib Dose in Patients with Advanced Breast Cancer with Renal Impairment Based on PK, Safety, and Efficacy Data: An Innovative Approach Integrating Data from a Dedicated Renal Impairment Study and Oncology Clinical Trials. Clin Pharmacokinet. 2023 Mar;62(3):493-504. doi: 10.1007/s40262-022-01206-2. Epub 2023 Feb 17. PMID 36800111